CLINICAL TRIAL: NCT06128980
Title: Withdrawal of Pharmacological Treatment for Heart Failure Patients With Recovery From Tachycardia-induced Cardiomyopathy - WEAN-HF
Brief Title: Withdrawal of Treatment for Heart Failure Patients With Recovery From Tachycardia-induced Cardiomyopathy
Acronym: WEAN-HF
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Collaborators: Nordsjaellands Hospital (Other); University Hospital Bispebjerg and Frederiksberg (Other); Zealand University Hospital (Other); Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Emil Wolsk, Head of Heart Failure, Principal investigator, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WEAN-HF
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Heart Failure With Reduced Ejection Fraction; Heart Rhythm Disorder

STUDY DESIGN:
Intervention Model Description: Randomized, non-inferiority study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Patients will be treated with GDMT for heart failure during the trial follow-up of 1 year.
- Weaning (Active Comparator): Patients will be weaned from GDMT in a sequential order.
  Interventions: Drug: GDMT

INTERVENTIONS:
Drug: GDMT — Sequential weaning starting with SGLT2i - MRA - BB - ACEi/ARB/ARNi
  Arms: Weaning

SUMMARY:
New onset heart failure (HF) is observed in up to 25% of patients with incident atrial fibrillation or flutter (AF). Current guidelines suggest that both conditions (AF & HF) be addressed with guideline directed medical therapy (GDMT) for HF and rate or rhythm control of AF. Hence, patients with both conditions are subjected to extensive polypharmacy with possible prognostic benefits, but also possible side effects, such as decreased renal function, dizziness, tiredness and hypotension, as well as the financial burden on both the individual patients and society, in addition to the stigma of having a HF diagnosis.

Guidelines do not inform how to manage long-term patients with HF, who following control of the incident tachycardia (e.g. AF), show full recovery from their HF condition.

This investigator-initiated, open-label, randomized, non-inferiority trial will test whether incremental weaning of GDMT in patients following full cardiac recovery and AF control is non-inferior compared to continuous GDMT with respect to the primary endpoint of freedom from heart failure deterioration. Furthermore, this study seeks to extensively phenotype these patients (genetic testing, advanced imaging, biomarkers etc.) in order to establish whether certain phenotypes are at lesser or greater risk of deterioration once remission is established. This novel approach of a personalized treatment regimen depending on e.g. genetic profiling could lead to an aggressive treatment in patients at high risk of deterioration and conversely spare patients with a negligible risk, a life-long intensive treatment regimen.

All HF clinics located in Zealand, Denmark, with a catchment area of >2 million citizens, have agreed to participate in the WEAN-HF trial. A total of 348 patients will be randomized. Patients are followed up the 1st year after randomization with clinical examination, biomarkers and echocardiography, and are subsequently followed via Danish nationwide registries for 10 years.

DETAILED DESCRIPTION:
Background:

Heart failure (HF) is a disease that affects more than 60000 patients in Denmark and millions across the world. The prognosis of HF is comparable to many types of cancer. New onset HF is observed in up to 25% of patients with incident atrial fibrillation or flutter (AF). The persistent tachycardia caused by AF is believed to exert the heart to a point where it causes HF. Whether AF is the cause of HF, or conversely that the detrimental effects of HF has induced AF, is difficult to ascertain upon the initial presentation. Current guidelines suggest that both conditions (AF & HF) be addressed with guideline directed medical therapy (GDMT) for HF and rate or rhythm control of AF. GDMT for HF consists of at least 4 different types of medication which is combined with management for AF (anticoagulant and often antiarrhythmic medication or ablation procedures). Hence, patients with both conditions are subjected to polypharmacy with at least 6 different types of medication in addition to their usual medication regimen. This may have prognostic benefits, but also possible side effects, such as decreased renal function, dizziness, tiredness and hypotension, as well as the financial burden on both the individual patients and society, in addition to the stigma of having a heart failure diagnosis.

Gaps in knowledge Data are lacking on how to optimally manage patients long-term with heart failure suspected to be tachycardia-induced, who following cessation or control of the incident AF, show full recovery from their heart failure condition. Guidelines do not suggest whether GDMT for heart failure should continue lifelong, cease or be weaned. In the TRED-HF study, 51 non-ischemic HF patients with LVEF recovery who were seemingly clinically stable were weaned from GDMT. Approximately 40% of patients showed signs of deterioration after 6 months of incremental GDMT weaning. Where TRED-HF patients had verified longstanding chronic HF, the situation for patients experiencing an incident episode of AF subsequently leading to acute heart failure may represent a different phenotype with a better prognosis once AF is terminated or controlled as suggested by observational data. Currently there is no data supporting how to manage GDMT in this population of heart failure patients with recovery following control of their AF episode.

Objective:

To observe whether incremental weaning of GDMT in patients following full cardiac recovery and AF control is non-inferior compared to continuous GDMT.

Furthermore, using an extensive phenotypic profiling, to investigate if one or more biomarkers can predict which patients are at an increased risk of cardiac deterioration in both intervention groups.

Hypothesis:

The investigators hypothesize that patients weaned from GDMT will experience similar rates of deterioration as patients on continuous GDMT.

Perspective The chance of remission after a heart failure diagnosis differs greatly depending on the etiology of heart failure. Although dramatic differences in remission rates depending on etiology have been established, patients with heart failure are in general committed to the same regimen of GDMT. For example, in patients with alcohol-induced heart failure, removing the cardiotoxic substance (alcohol) through abstinence leads to recovery in >50% of cases. Genetic profiling reveals that changes in mutations leading to alterations in cardiac structural proteins - titin - are very prevalent in patients with alcohol-induced heart failure. It appears that patients may be at increased risk of heart failure if they both have a genetic disposition combined with a cardiotoxic stimulus (e.g. alcohol, tachycardia). Interestingly, mutations in the same titin gene has also been found in many patients with atrial fibrillation. Therefore, it is plausible that if the detrimental effects of prolonged tachycardia could be stopped a continuous HF remission in our cohort would be observed. This study seeks to extensively phenotype patients with tachycardia-induced heart failure in order to establish whether certain phenotypes are at lesser or greater risk of deterioration once remission is established. This novel approach of a personalized heart failure treatment regimen depending on genetic profiling and advanced imaging could lead to an aggressive treatment in patients at high risk of deterioration and conversely spare patients with a negligible risk of deterioration a life-long intensive treatment regimen.

Primary endpoint:

Patients free from heart failure deterioration 1 year after randomization

Secondary endpoints 1 year after randomization:

* Changes in Minnesota Living with Heart Failure Questionnaire from baseline (min. score 0 - max. score 105, where higher scores indicates worse quality of life)
* Hospitalization for heart failure
* Cardiovascular (CV) hospitalizations
* Non-CV hospitalizations
* CV death
* All-cause death
* Patients in need of initiation of loop diuretics or doubling of dosage
* Changes in N-terminal pro-Brain Natriuretic Peptide (NT-proBNP) from baseline
* Patients needing changes in medication for AF (uptitration of current medication or change in/addition of new medication) or re-do ablation for AF
* Patients with signs of AF that persistently exceed 110 bpm despite best practice Adverse events will be summarized;
* Patients with renal deterioration, hypotension, dizziness.
* Patients with signs of new onset liver affection and/or thyroid dysfunction

Methods:

This is an investigator-initiated, open-label, randomized, non-inferiority trial. This clinical trial complies with the Declaration of Helsinki, modified in 2013. This study has been approved by both the ethical committee (H-23010220) and the Knowledge Centre on Data Protection Compliance in the Capital Region of Denmark (P-2023-111). This trial will adhere to good clinical practice guidelines (GCP).

Patients with HF who are followed in HF clinics on Zealand including the greater Copenhagen region are screened. This area covers >2 million citizens (approximately 1/3 of all citizens in Denmark). All patients fulfilling criteria for participation will be invited to participate. HF specialists at each HF clinic will assess eligibility based on a review of the medical chart and an individual assessment. Patients can be rescreened for inclusion repeatedly throughout the inclusion period.

Collaborators:

This trial is executed, analyzed and published by the main applicant and nested at Herlev-Gentofte Hospital. A collaboration between the applicant and heart failure clinics is pivotal in order to ensure timely inclusion of a generalizable heart failure population and to swiftly implement the findings into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Patients with new onset heart failure (ambulatory or hospital) with reduced ejection fraction (LVEF≤40% assessed by echocardiography) and NYHA ≥2 and atrial fibrillation or atrial flutter with ventricular rate ≥110 bpm (ECG monitoring, hospital telemetry or Holter monitoring) that following GDMT - while AF is terminated (e.g. ablation or conversion) or controlled (HR<110 on resting ECG) - experience LVEF remission (LVEF ≥50%), normalization of indexed LV volume, and normal ECG (no bundle branch block, ST segment deviations or T-wave inversion) within 3 months after GDMT.

Exclusion Criteria:

* 18 years or older and able to consent
* Former ablation procedures and inability to tolerate antiarrhythmic drugs
* Pregnancy
* Congenital heart disease (congenital defects with no hemodyamic effects are not excluded)
* Previously genotyped positive for genes known to cause cardiomyopathy
* Probable hypertrophic, restrictive or non-compaction cardiomyopathy
* Moderate/severe valvular disease
* Suspicion of or known cardiac amyloidosis, sarcoidosis, or other storage/inflammatory disease
* More than 10% PVCs or documented sustained ventricular arrhythmias
* History of persistent or permanent AF with ventricular rates >110 before incident HF despite best standard of care
* eGFR < 40 ml/min/1.73 m2
* Acute myocardial infarction at index
* Probable medication-, alcohol- or illicit drug use induced AF and/or HF
* Systolic blood pressure >160 mmHg (at multiple measurements) at index or history of uncontrollable hypertension
* Myocarditis
* Cardiogenic shock at index
* Aborted sudden cardiac death
* Pacing-induced cardiomyopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Patients free from heart failure deterioration 1 year after randomization | 1 year after randomization
  Heart failure deterioration is defined as following; a reduction in LVEF of more than 10% and less than 50%, and/or increase in LVEDV by more than 10% and to higher than the normal range (indexed for body surface area), and/or hospitalization for heart failure and/or arrhythmia, and/or clinical evidence of heart failure.

SECONDARY OUTCOMES:
Changes in Minnesota Living with Heart Failure Questionnaire from baseline | 1 year after randomization
  Between group changes will be analysed
Hospitalization for heart failure | 1 year after randomization
  Time to 1st and total HF hospitalizations
Cardiovascular (CV) hospitalizations | 1 year after randomization
  Time to 1st and total CV hospitalizations
Non-CV hospitalizations | 1 year after randomization + 10 year follow-up
  Time to 1st and total non-CV hospitalizations
CV death | 1 year after randomization + 10 year follow-up
  Incidence rates with between group comparisons
All-cause death | 1 year after randomization + 10 year follow-up
  Incidence rates with between group comparisons
Patients in need of initiation of loop diuretics or doubling of dosage | 1 year after randomization
  Incidence rates with between group comparisons
Changes in N-terminal pro-Brain Natriuretic Peptide (NT-proBNP) from baseline | 1 year after randomization
  Between group comparisons
Patients needing changes in medication for AF (uptitration of current medication or change in/addition of new medication) or re-do ablation for AF | 1 year after randomization
  Between group comparisons
Patients with signs of AF that persistently exceed 110 bpm despite best practice | 1 year after randomization
  Between group comparisons

OTHER OUTCOMES:
Patients with renal deterioration, hypotension, dizziness. | 1 year after randomization
  Between group comparisons
Patients with signs of new onset liver affection and/or thyroid dysfunction | 1 year after randomization
  Between group comparisons

CONTACTS AND LOCATIONS:
Overall Officials: Emil Wolsk, MD, Principal Investigator — Herlev and Gentofte Hospital
Locations (1):
- Herlev-Gentofte Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No